CLINICAL TRIAL: NCT06082115
Title: Functional Outcome of Mirror Therapy Versus Task Oriented Training on Hand Function in Children With Unilateral Cerebral Palsy
Brief Title: Mirror Therapy Versus Task Oriented Training on Hand Function in Children With Unilateral Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Eman Wagdy, Lecturer, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004452
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Unilateral Cerebral Palsy
Keywords: Mirror Therapy; Task Oriented Training; Hand Function; Unilateral Cerebral Palsy
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Selected Physical Therapy Program, Mirror Therapy, Task Oriented Training
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Selected Physical and Occupational Therapy Program (Experimental): Unilateral cerebral palsy children will receive selected physical and occupational therapy program for 1 hour. The duration of treatment will be 3 times/week for 12 weeks.
  Interventions: Other: Selected Physical and Occupational Therapy Program
- Mirror Therapy (Experimental): Unilateral cerebral palsy children will receive selected physical and occupational therapy program for 1 hour in addition to mirror therapy for 30 minutes. The duration of treatment will be 3 times/week for 12 weeks.
  Interventions: Other: Selected Physical and Occupational Therapy Program; Other: Mirror Therapy
- Task Oriented Training (Experimental): Unilateral cerebral palsy children will receive selected physical and occupational therapy program for 1 hour in addition to task oriented training for 30 minutes. The duration of treatment will be 3 times/week for 12 weeks.
  Interventions: Other: Selected Physical and Occupational Therapy Program; Other: Task-Oriented Training

INTERVENTIONS:
Other: Selected Physical and Occupational Therapy Program — The selected physical and occupational therapy program include:- A-Physical therapy program contains neurodevelopmental technique for U.L & L.L (U.L & L.L approximation, U.L & L.L weight bearing exercises), stretching exercises for U.L & L.L muscles, strengthening exercises for antispastic group of U.L & L.L muscles, facilitation of postural reactions, facilitation of gait training and, ascending and descending stairs.
  B-Occupational therapy program contains transfer cube from one hand to hand, reaching to mouth (eating lollipop), throwing and catching ball and, clapping with both hands.
Other: Mirror Therapy — The mirror therapy program include tasks of manipulative and grasping skills that performed by the non-affected hand in-front of mirror while the affected hand behind the mirror. These tasks contain building towers, rolling dough, transferring cup from one place to another place, turning cards, moving keys, drawing circle and, grasps various objects with different size, shape and weight (ball, markers, pegs and brushes).
  Arms: Mirror Therapy
Other: Task-Oriented Training — The task-oriented training program include tasks of manipulative and grasping skills that performed by the affected hand based on repetition practice. These tasks contain building towers, rolling dough, transferring cup from one place to another place, turning cards, moving keys, drawing circle and, grasps various objects with different size, shape and weight (ball, markers, pegs and brushes).
  Arms: Task Oriented Training

SUMMARY:
The purpose of the study is to compare the effect between mirror therapy and task-oriented training on hand function in children with unilateral cerebral palsy.

DETAILED DESCRIPTION:
Dysfunction in the upper limbs and hand function is one of the most common symptoms in children with cerebral palsy (CP), particularly children with unilateral CP which intern has the potential to limit the involvement of these children in life activities and cause distress and suffering for both children and their parents. Different rehabilitation intervention procedures addressing upper extremity dysfunction are essential to promote better use of disabled arms and hands in daily activities and achieving functional independence at home, in school and in the community. However, there is little evidence directed toward which intervention procedure is more effective on hand function therefore, there is need to compare between the functional outcome of mirror therapy versus task-oriented training on hand function in children with unilateral cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages will be ranged from 5 to 8 years old.
2. Wrist flexor spasticity ranged from grade 1 to 1+ according to Modified Aswarth scale.
3. Capacity to handle objects without continuous assistance (level I or II in accordance with the Manual Ability Classification System).
4. Ability to sit alone.
5. Sufficient cognition to follow simple verbal instructions.

Exclusion Criteria:

1. Fixed contracture or deformities in the upper limb.
2. Visual or auditory defects.
3. Botulinuim toxin injection in the last 6 months before the study.
4. Previous surgical intervention in the upper limb.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | Up to 12 weeks
  Hand-held dynamometer will be used to measure hand grip strength. It is a valid and reliable device used to measure isometric grip strength.

SECONDARY OUTCOMES:
Range of Motion | Up to 12 weeks
  Electronic(digital) goniometer will be used for measuring wrist extension ROM. It is a valid and reliable tool used to assess wrist extension ROM
Upper Extremity Skills | Up to 12 weeks
  Quality Upper Extremity Skill Test (QUEST) will be used to evaluate movement pattern and and function. It is a valid scale contains 4 domains (33 items); Dissociated movements (19 items), Grasp (6 items), Weight bearing (5 items) and Protective extension (3 items). The total testing time including administration and scoring is approximately 45 minutes.
Hand Dexetrity | Up to 12 weeks
  Box and Block Test (BBT) will be used for measuring hand dexterity by using two compartment box containing 150 blocks. The test includes grasping, moving, and releasing wooden blocks from one side to the other. The score was recorded for 1 minute as the number of blocks passed over the wooden partition